CLINICAL TRIAL: NCT01489644
Title: A Randomized, Single-Blind, Four-Period Crossover Study Examining the Single Dose Pharmacokinetics of Repaglinide, Metformin and Combination Tablet Dosing (NN4440) in Fasting and Fed Healthy Volunteers
Brief Title: Single Dose Pharmacokinetics of Repaglinide, Metformin and Combination Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NN4440-1779
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment period 1 (Experimental)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet
- Treatment period 2 (Experimental)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet
- Treatment period 3 (Experimental)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet
- Treatment period 4 (Active Comparator)
  Interventions: Drug: repaglinide; Drug: metformin; Drug: repaglinide and metformin combination tablet

INTERVENTIONS:
Drug: repaglinide — Subjects will receive 850 mg metformin alone on a fasting state, 2 mg repaglinide alone on a fasting state, 2 mg repaglinide/850 mg metformin (NN4440 2/850) in the fasting state or 2 mg repaglinide/850 mg metformin (NN4440 2/850) immediately prior to a standardised high fat meal on 4 separate dosing visits in varying order
Drug: metformin — Subjects will receive 850 mg metformin alone on a fasting state, 2 mg repaglinide alone on a fasting state, 2 mg repaglinide/850 mg metformin (NN4440 2/850) in the fasting state or 2 mg repaglinide/850 mg metformin (NN4440 2/850) immediately prior to a standardised high fat meal on 4 separate dosing visits in varying order
Drug: repaglinide and metformin combination tablet — Subjects will receive 850 mg metformin alone on a fasting state, 2 mg repaglinide alone on a fasting state, 2 mg repaglinide/850 mg metformin (NN4440 2/850) in the fasting state or 2 mg repaglinide/850 mg metformin (NN4440 2/850) immediately prior to a standardised high fat meal on 4 separate dosing visits in varying order

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare repaglinide and metformin administered as an individual tablets with repaglinide and metformin administered as a combination tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers (female not pregnant, lactating or breastfeeding)
* BMI (Body Mass Index) between 19-29 kg/m^2, both inclusive
* Fasting plasma glucose from 70-115 mg/dl
* Subject is judged to be in good health on the basis of their medical history, physical examination, ECG (electrocardiogram), and routine laboratory data

Exclusion Criteria:

* Any clinically significant disease history, in the opinion of the Investigator, of systemic or organ disease
* Clinically significant abnormalities on pre-study clinical examination or any laboratory measurements during screening
* Positive results on Screening for Hepatitis B surface antigen, Hepatitis C antibody and HIV (human immunodeficiency virus) antibody
* Positive results on the drug abuse/alcohol screen
* Any regular use of prescription or nonprescription drugs, including mega-vitamin, health food or dietary supplement regimens, with the exception of contraceptives, that cannot be stopped at least 1 week prior to Visit 2 (trial product administration) and for the duration of the study
* Subject is currently a smoker (more than one cigarette per day or equivalent)
* Use of grapefruit or grapefruit juice within 7 days of trial product administration
* Blood donation, surgery or trauma with significant blood loss (500 mL) within the last 2 months prior to dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Fasting repaglinide and metformin Area under the Curve (AUC) following NN4440 administration
Fasting repaglinide and metformin Area under the Curve (AUC) following individual administration
Fasting repaglinide and metformin Cmax (maximum drug concentration) following NN4440 administration
Fasting repaglinide and metformin Cmax (maximum drug concentration) following individual administration

SECONDARY OUTCOMES:
Repaglinide and metformin tmax (time to maximum) following individual administration fasting state
Repaglinide and metformin tmax (time to maximum) following NN4440 administration fasting state
Physical examinations
Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Tacoma, Washington

REFERENCES:
- [Result] Reilley S, Chang C-T, Lyness W. Single-Dose Pharmacokinetics of a Repaglinide/Metformin Fixed-Dose Combination Tablet in Fasted and Fed Conditions. Diabetes 2008; 57 (Suppl 1): 2449 in 01-D
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com